CLINICAL TRIAL: NCT01792804
Title: Early Oral Switch Therapy in Low-risk Staphylococcus Aureus Bloodstream Infection
Brief Title: Staphylococcus Aureus Bacteremia Antibiotic Treatment Options
Acronym: SABATO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-1400; 2013-000577-77 (EudraCT Number)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Staphylococcus Aureus Infection
Keywords: Staphylococcus aureus; Bloodstream infection; Oral switch
MeSH Terms: conditions — Staphylococcal Infections; Sepsis | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Clindamycin; Linezolid; Floxacillin; Cloxacillin; Vancomycin; Daptomycin; Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orally administered antibiotic (Experimental): First choice (MRSA and MSSA): trimethoprim-sulfamethoxazole, or Second choice (MSSA): clindamycin, or Second choice (MRSA): linezolid administered for 7-9 days
  Interventions: Drug: Trimethoprim-Sulfamethoxazole; Drug: Clindamycin; Drug: Linezolid
- Intravenously administered antibiotic (Experimental): First choice (MSSA): flucloxacillin [Spain: cloxacillin], or cefazolin or Second choice (MSSA): vancomycin, or First choice (MRSA): vancomycin, or Second choice (MRSA): daptomycin administered for 7-9 days
  Interventions: Drug: Flucloxacillin; Drug: Cloxacillin; Drug: Vancomycin; Drug: Daptomycin; Drug: Cefazolin

INTERVENTIONS:
Drug: Trimethoprim-Sulfamethoxazole — study drug 1
  Arms: Orally administered antibiotic
Drug: Clindamycin — study drug 2
  Arms: Orally administered antibiotic
Drug: Linezolid — study drug 3
  Arms: Orally administered antibiotic
Drug: Flucloxacillin — study drug 4
  Arms: Intravenously administered antibiotic
Drug: Cloxacillin — study drug 5
  Arms: Intravenously administered antibiotic
Drug: Vancomycin — study drug 6
  Arms: Intravenously administered antibiotic
Drug: Daptomycin — study drug 7
  Arms: Intravenously administered antibiotic
Drug: Cefazolin — study drug 8
  Arms: Intravenously administered antibiotic

SUMMARY:
Increasing resistance to antibiotic agents has been recognized as a major health problem worldwide that will even aggravate due to the lack of new antimicrobial agents within the next decade [1]. This threat underscores the need to maximize clinical utility of existing antibiotics, through more rational prescription, e.g. optimizing duration of treatment.

Staphylococcus aureus bloodstream infection (SAB) is a common disease with about 200,000 cases occurring annually in Europe [2]. A course of at least 14 days of intravenous antimicrobials is considered standard therapy [3-5] in "uncomplicated" SAB. This relatively long course serves to prevent SAB-related complications (such as endocarditis and vertebral osteomyelitis) that may result from hematogenous dissemination to distant sites. However, there is insufficient evidence that a full course of intravenous antibiotic therapy is always required in patients with a low risk of SAB-related complications.

In a multicenter, open-label, randomized controlled trial we aim to demonstrate that an early switch from intravenous to oral antimicrobial therapy is non-inferior to a conventional 14-days course of intravenous therapy regarding efficacy and safety. An early switch from intravenous to oral therapy would provide several benefits such as earlier discharge, fewer adverse reactions associated with intravenous therapy, increased quality of life, and cost savings.

DETAILED DESCRIPTION:
1. WHO. WHO Global Strategy for Containment of Antimicrobial Resistance.: World Health Organization, 2001.
2. Kern WV. Management of Staphylococcus aureus bacteremia and endocarditis: progresses and challenges. Curr Opin Infect Dis 2010;23(4):346-58.
3. Gemmell CG, Edwards DI, Fraise AP, Gould FK, Ridgway GL, Warren RE. Guidelines for the prophylaxis and treatment of methicillin-resistant Staphylococcus aureus (MRSA) infections in the UK. J Antimicrob Chemother 2006;57(4):589-608.
4. Liu C, Bayer A, Cosgrove SE, et al. Clinical practice guidelines by the Infectious Diseases Society of America for the treatment of methicillin-resistant Staphylococcus aureus infections in adults and children. Clin Infect Dis 2011;52(3):e18-55.
5. Mermel LA, Allon M, Bouza E, et al. Clinical practice guidelines for the diagnosis and management of intravascular catheter-related infection: 2009 Update by the Infectious Diseases Society of America. Clin Infect Dis 2009;49(1):1-45.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Not legally incapacitated
* Written informed consent from the trial subject has been obtained
* Blood culture positive for S. aureus not considered to represent contamination
* At least one negative follow-up blood culture obtained within 24-96 hours after the start of adequate antimicrobial therapy to rule out persistent bacteremia and Absence of a blood culture positive for S. aureus at the same time or thereafter.
* Five to seven full days of appropriate i.v. antimicrobial therapy administered prior to randomization documented in the patient Chart. Appropriate therapy has all of the following characteristics:

  1. Antimicrobial therapy has to be initiated within 72h after the first positive blood culture was drawn.
  2. Provided in-vitro susceptibility and adequate dosing (as judged by the PI) preferred agents for pre-randomization antimicrobial therapy are flucloxacillin, cloxacillin, vancomycin and daptomycin. However, the following antimicrobials are allowed:

     * MSSR: penicillinase-resistant penicillins (e.g. flucloxacillin, cloxacillin), β-lactam plus β-lactamase-inhibitors (e.g. ampicillin+sulbactam, piperacillin+tazobactam), cephalosporins (except ceftazidime), carbapenems, clindamycin, fluoroquinolones, trimethoprimsulfamethoxazole, doxycycline, tigecycline, vancomycin, teicoplanin, telavancin, linezolid, daptomycin, ceftaroline, ceftobiprole, and macrolides.
     * MRSA: vancomycin, teicoplanin, telavancin, fluoroquinolones, clindamycin, trimethoprim-sulfamethoxazole, doxycycline, tigecycline, linezolid, daptomycin, macrolides, ceftaroline, and ceftobiprole.

Exclusion Criteria:

* Polymicrobial bloodstream infection, defined as isolation of pathogens other than S. aureus from a blood culture obtained in the time from two days prior to the first positive blood culture with S. aureus until randomization. Common skin contaminants (coagulase-negative staphylococci, diphtheroids, Bacillus spp., and Propionibacterium spp.) detected in one of several blood cultures will not be considered to represent polymicrobial infection
* Recent history (within 3 months) of prior S. aureus bloodstream infection
* In vitro resistance of S. aureus to all oral or all i.v. study drugs
* Contraindications for all oral or all i.v. study drugs
* Previously planned Treatment with active drug against S. aureus during Intervention Phase (e.g. cotrimoxazol prophylaxis)
* Signs and symptoms of complicated SAB as judged by an ID physician. Complicated infection is defined as at least one of the following:

  * deep-seated focus: e.g. endocarditis, pneumonia, undrained abscess, empyema, and Osteomyelitis
  * septic shock, as defined by the AACP criteria (23), within 4 days before randomization
  * prolonged bacteremia: positive follow-up blood culture more than 72h after the start of adequate antimicrobial therapy
  * body temperature >38 °C on two separate days within 48h before randomization
* Presence of the following non-removable foreign bodies (if not removed 2 days or more before randomization):

  * prosthetic heart valve
  * deep-seated vascular graft with foreign material (e.g. PTFE or dacron graft). Hemodialysis shunts are not considered deep-seated vascular grafts.
  * ventriculo-atrial shunt
* Presence of a prosthetic joint (if not removed 2 days or more before randomization). This is not an exclusion criterion, if all of the following conditions are fulfilled:

  * prosthetic joint was implanted at least 6 months prior, and
  * catheter-related infection, skin and soft tissue infection, or surgical wound infection is present (as defined below), and
  * joint infection unlikely (no clinical or imaging signs)
* Presence of a pacemaker or an automated implantable cardioverter Defibrillator (AICD) device (if not removed 2 days or more before randomization). This is not an exclusion criterion, if all of the following conditions are fulfilled:

  * pacemaker or AICD was implanted at least 6 months prior, and
  * catheter-related infection, skin and soft tissue infection, or surgical wound infection is present (as defined below), and
  * no clinical signs of infective endocarditis, and
  * infective endocarditis unlikely by echocardiography (preferably TEE), and
  * pocket infection unlikely (no clinical or imaging signs)
* Failure to remove any intravascular catheter which was present when first positive blood culture was drawn within 4 days of the first positive blood culture
* Severe liver disease. This is not an exclusion criterion, if the following condition is fulfilled:

  - catheter-related infection, skin and soft tissue infection, or surgical wound infection is present
* End-stage renal disease. This is not an exclusion criterion, if all of the following conditions are fulfilled:

  * catheter-related infection, skin and soft tissue infection, or surgical wound infection is present (as defined below), and
  * no clinical signs of infective endocarditis, and
  * infective endocarditis unlikely by echocardiography (preferably TEE), and
  * in patients with a hemodialysis shunt with a non-removable foreign body (e.g. synthetic PTFE loop): no clinical signs of a shunt infection
* Severe immunodeficiency

  * primary immunodeficiency disorders
  * neutropenia (<500 neutrophils/μl) at randomization or neutropenia expected during intervention phase due to immunosuppressive treatment
  * uncontrolled disease in HIV-positive patients
  * high-dose steroid therapy (>1 mg/kg prednisone or equivalent doses given for >4 weeks or planned during intervention)
  * immunosuppressive combination therapy with two or more drugs with different mode of action
  * hematopoietic stem cell transplantation within the past 6 months or planned during treatment period
  * solid organ transplant
  * treatment with biologicals within the previous year
* Life expectancy < 3 months
* Inability to take oral drugs
* Injection drug user
* Expected low compliance with drug regimen
* Participation in other interventional trials within the previous three months or ongoing
* Pregnant women and nursing mothers
* For premenopausal women: Failure to use highly-effective contraceptive methods for 1 month after receiving study drug. The following contraceptive methods with a Pearl Index lower than 1% are regarded as highly-effective:

  * oral hormonal contraception ('pill')
  * dermal hormonal contraception
  * vaginal hormonal contraception (NuvaRing®)
  * contraceptive plaster
  * long-acting injectable contraceptives
  * implants that release progesterone (Implanon®)
  * tubal ligation (female sterilisation)
  * intrauterine devices that release hormones (hormone spiral)
  * double barrier methods
* Persons with any kind of dependency on the investigator or employed by the sponsor or investigator
* Persons held in an institution by legal or official order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
SAB-related complications | 90 days
  S. aureus bloodstream infection-related complications (relapsing SAB, deep-seated infection with S. aureus, or attributable mortality) within 90 days

SECONDARY OUTCOMES:
Length of hospital stay | 90 days
  Length of hospital stay
Survival | 14, 30, and 90 days
  Survival at 14, 30, and 90 days
Complications of intravenous therapy | 90 days
  Complications of intravenous therapy, such as thrombophlebitis.

OTHER OUTCOMES:
Clostridium difficile associated diarrhea (CDAD) | 90 days
  Clostridium difficile associated diarrhea (CDAD)
AEs and SAEs | 90 days
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Achim J Kaasch, MD, Principal Investigator — Heinrich-Heine University, Duesseldorf
Locations (40):
- France (15):
  - Annecy, Annecy
  - Chambéry, Chambéry
  - Grenoble, Grenoble
  - La Roche-sur-Yon, La Roche-sur-Yon
  - Nantes, Nantes
  - Orléans, Orléans
  - Paris 5, Paris
  - Paris 1, Paris
  - Paris 3, Paris
  - Paris 2, Paris
  - Paris 4, Paris
  - Quimper, Quimper
  - Rennes, Rennes
  - St. Etienne, Saint-Etienne
  - Tours, Tours
- Germany (11):
  - Berlin, Berlin
  - Uniklinik Köln, Cologne
  - Düsseldorf, Düsseldorf
  - Frankfurt, Frankfurt am Main
  - Freiburg, Freiburg im Breisgau
  - Hannover, Hanover
  - Jena, Jena
  - Krefeld, Krefeld
  - Leverkusen, Leverkusen
  - Lübeck, Lübeck
  - Ulm, Ulm
- Netherlands (8):
  - VUmc Amsterdam, Amsterdam
  - Amsterdam, Amsterdam
  - Breda, Breda
  - Groningen, Groningen
  - UMC Groningen, Groningen
  - Tilburg, Tilburg
  - Utrecht, Utrecht
  - Diakonessenhuis Utrecht, Utrecht
- Spain (5):
  - Barcelona II, Barcelona
  - Barcelona I, Barcelona
  - Palma, Palma de Mallorca
  - Sevilla II, Seville
  - Sevilla, Seville
- Nottingham, Nottingham, United Kingdom

REFERENCES:
- [Derived] Kaasch AJ, Lopez-Cortes LE, Rodriguez-Bano J, Cisneros JM, Dolores Navarro M, Fatkenheuer G, Jung N, Rieg S, Lepeule R, Coutte L, Bernard L, Lemaignen A, Kosters K, MacKenzie CR, Soriano A, Hagel S, Fantin B, Lafaurie M, Talarmin JP, Dinh A, Guimard T, Boutoille D, Welte T, Reuter S, Kluytmans J, Martin ML, Forestier E, Stocker H, Vitrat V, Tattevin P, Rommerskirchen A, Noret M, Adams A, Kern WV, Hellmich M, Seifert H; SABATO study group. Efficacy and safety of an early oral switch in low-risk Staphylococcus aureus bloodstream infection (SABATO): an international, open-label, parallel-group, randomised, controlled, non-inferiority trial. Lancet Infect Dis. 2024 May;24(5):523-534. doi: 10.1016/S1473-3099(23)00756-9. Epub 2024 Jan 17. PMID 38244557
- [Derived] Kaasch AJ, Rommerskirchen A, Hellmich M, Fatkenheuer G, Prinz-Langenohl R, Rieg S, Kern WV, Seifert H; SABATO trial group. Protocol update for the SABATO trial: a randomized controlled trial to assess early oral switch therapy in low-risk Staphylococcus aureus bloodstream infection. Trials. 2020 Feb 12;21(1):175. doi: 10.1186/s13063-020-4102-0. PMID 32051007
- [Derived] Kaasch AJ, Fatkenheuer G, Prinz-Langenohl R, Paulus U, Hellmich M, Weiss V, Jung N, Rieg S, Kern WV, Seifert H; SABATO trial group (with linked authorship to the individuals in the Acknowledgements section). Early oral switch therapy in low-risk Staphylococcus aureus bloodstream infection (SABATO): study protocol for a randomized controlled trial. Trials. 2015 Oct 9;16:450. doi: 10.1186/s13063-015-0973-x. PMID 26452342